CLINICAL TRIAL: NCT04839445
Title: Comparison of Efficacy of Ultrasound-guided Erector Spinae Place Block Versus Transversus Abdominis Plane Block for Intra and Postoperative Pain Control in Total Laparoscopic Hysterectomy: a Randomized Controlled Trial
Brief Title: ESP vs TAP in Total Laparoscopic Hysterectomy
Acronym: ARTEMIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AUSL Romagna Rimini (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2909
Record Dates: First submitted 2021-04-05; First posted 2021-04-09 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-04

CONDITIONS: Anesthesia; Gynecologic Cancer
Keywords: Transversus Abdominal Plane Block; Erector Spinae Plane Block; General Anesthesia; Laparoscopic Hysterectomy
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia + TAP block (Active Comparator): Induction: remifentanil in total intravenous anesthesia (TIVA), Propofol 2 mg/kg/h and Rocuronium 0.6 mg/kg. Transversus abdominis plane (TAP) block: 20 minutes before surgery. Ropivacaine 0.37% 20ml + dexamethasone 2mg per side. Maintenance: TIVA with Propofol, the infusion rate will be adjusted according to the bispectral index system (BIS) values (30 <BIS <50). Patients will receive additional remifentanil by infusion at 0.02 mcg/kg/min per time if blood pressure and heart rate values exceed 20% pre-operative baseline values. Additional rocuronium 0.1 mg/kg based on clinical needs and train of four (TOF) monitoring. Analgesic starter bolus: 30 minutes before the end of the surgery, paracetamol 1 gr ev and ketorolac 30 mg ev. Postoperative pain: paracetamol 1 gr ev every 8 hours for 36 hours; ketorolac 30 mg ev if NRS >4 / morphine 2 mg ev if NRS >4 30 min after ketorolac administration. In case of nausea and vomiting ondansetron 4 mg ev.
  Interventions: Procedure: General anesthesia + TAP block
- General anesthesia + ESP block (Active Comparator): Erector spinae plane (ESP) block: 20 minutes before surgery. T8 level bilaterally, ropivacaine 0.37% 20ml + dexamethasone 2mg per side.
  Induction: Remifentanil in TIVA, Propofol 2 mg/kg/h and Rocuronium 0.6 mg/kg. Maintenance: TIVA with Propofol, the infusion rate will be adjusted according to the BIS values (30 <BIS <50). Patients will receive additional remifentanil by infusion at 0.02 mcg/kg/min per time if blood pressure and heart rate values exceed 20% pre-operative baseline values. Additional rocuronium 0.1 mg/kg based on clinical needs and TOF monitoring.
  Analgesic starter bolus: 30 minutes before the end of the surgery, paracetamol 1 gr ev and ketorolac 30 mg ev.
  Postoperative pain: paracetamol 1 gr ev every 8 hours for 36 hours; ketorolac 30 mg ev if NRS >4 / morphine 2 mg ev if NRS >4 30 min after ketorolac administration. In case of nausea and vomiting ondansetron 4 mg ev.
  Interventions: Procedure: General anesthesia + ESP block

INTERVENTIONS:
Procedure: General anesthesia + TAP block — Post induction TAP block for intra and postoperative analgesia.
  Arms: General anesthesia + TAP block
Procedure: General anesthesia + ESP block — Pre induction ESP block for intra and postoperative analgesia.
  Arms: General anesthesia + ESP block

SUMMARY:
The anesthetic techniques for videolaparoscopic surgery include general anesthesia, and locoregional anesthesia in association with general anesthesia in order to reduce or abolish post-operative pain with a simultaneous reduction in the use of opioids and days of hospital stay.

From the studies published so far on videolaparoscopic surgery in general, it is clear that the transversus abdominal plane (TAP) block could have a role in reducing the stretch wall pain secondary to pneumoperitoneum and incisional, although its role in this regard is not yet clear, nor significant statistically results have been produced. The use of erector spinae plane (ESP) block for the management of visceral pain is finding more and more space in the literature, with promising results.

For videolaparoscopic gynecological surgery, the techniques of locoregional anesthesia studied in association with general anesthesia, up to now, include wall blocks, TAP block and ESP block, while neuraxial anesthesia has no indications in this regard.

Although videolaparoscopic hysterectomy is considered less painful than the open-abdomen technique, it requires careful management of post-operative pain. The pain of this surgery is the result of the sum of incisional pain, at the insertion points of the laparoscopic trocars, pain due to pneumoperitoneum usually referred to the shoulder, and visceral pain purely dependent on surgical maneuvers. There is currently no strong evidence to support the use of locoregional anesthesia techniques in videolaparoscopic gynecological surgery. Few studies have been produced about this topic, and they are mostly case series or randomized controlled trials that take into consideration only one technique among those possible. To date, no study compares the various techniques to evaluate the possible superiority of one over the other.

In our hospital anesthesists carry out, in normal clinical practice, all the aforementioned local anesthesia techniques.

The purpose of our work is to evaluate, with a randomized non-sponsored study, the efficacy of the ESP block and the TAP block for intra and post-operative pain control in videolaparoscopic hysterectomy, and to compare the two techniques.

Based on the evidence available in the literature, the two techniques are already part of the current clinical practice of the Anesthesia Unit of our hospital and the choice of one technique over the other is based on anesthetist clinical evaluation to date. The anesthetists involved in the study are adequately trained on both anesthetic procedures.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists (ASA) I-III risk
* no contraindication to the execution of the peripheral nerve block
* signature of the informed consent
* total videolaparoscopic surgery (no conversion to open-abdomen)

Exclusion Criteria:

* allergies and / or contraindications to the administration of the drugs used in the study
* infections and injuries at the puncture site
* BMI ≥40
* history of opioid abuse or use of opioids in chronic therapy

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Postoperative pain control | 12 hours
  Evaluate the difference between the two groups regarding post-operative pain using Numeric Rating Scale (NRS) 0= better outcome; 10=worse outcome Score will be measured on the numeric rating scale (NRS), an NRS ≤ 4 will be considered as effective antalgic coverage.

SECONDARY OUTCOMES:
Intra operative use of opioids. | Surgery time.
  Mcg of Remifentanil consumed during surgery.
Post operative use of non-steroidal anti-inflammatory drugs | 2-6-12-24-36 postoperative hours
  Mg of ketorolac or any others anti-inflammatory drugs administered after surgery.
Post operative use of opioids | 2-6-12-24-36 postoperative hours
  Mg of opioids administered after surgery.
Postoperative nausea and / or vomiting | 2-6-12-24-36 postoperative hours
  Quantity of antiemetic drugs required to control nausea and vomiting episodes
Days of hospital stay | 3 days
  The number of days of hospitalization after surgery will be assessed
Assessment of patient satisfaction with the anesthesiological technique | 36 hours
  Patients is requested to fill out a pre-printed sheet on their judgment of the anesthesiological procedure, in which they can express a value from 0 to 5, where 0 indicates "entirely dissatisfied" and 5 indi- cates "very satisfied"expressed by the patient according to the following scale: satisfied, very satisfied, not at all satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Rosato, MD, Principal Investigator — AUSL Romagna
Locations (1):
- AUSL Romagna M. Bufalini Hospital, Cesena, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jones JH, Aldwinckle R. Interfascial Plane Blocks and Laparoscopic Abdominal Surgery: A Narrative Review. Local Reg Anesth. 2020 Oct 23;13:159-169. doi: 10.2147/LRA.S272694. eCollection 2020. PMID 33122942
- [Result] Bagaphou CT, Santonastaso DP, Rispoli M, Piraccini E, Fusco P, Gori F. Bilateral continuous erector spinae plane block: an alternative to epidural catheter for major open abdominal surgery. Minerva Anestesiol. 2020 Sep;86(9):993-994. doi: 10.23736/S0375-9393.20.14557-7. Epub 2020 Jun 2. No abstract available. PMID 32490608